CLINICAL TRIAL: NCT02176239
Title: Monitoring of 5% Treatment Naïve Intravenous Immunoglobulin (IVIg) Primary Immunodeficiency Disease (PIDD) Patients Using the CareExchange® System: A Pilot Study Using 5% Gammaplex® IVIg in the Home Setting
Status: Completed | Type: Observational
Sponsor: BriovaRx Infusion Services (Industry)
Collaborators: Bio Products Laboratory (BPL) (Unknown)
Responsible Party: Sponsor
Other Study IDs: AHS1-13-003
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Primary Immunodeficiency Disease (PIDD)
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gammaplex® IVIg

SUMMARY:
The purpose of this study is to demonstrate the utility of measuring outcomes in 5% treatment naïve Intravenous Immunoglobulin (IVIg) Primary Immunodeficiency Disease (PIDD) patients using infusion nurse and patient measured physical, quality of life (QOL), respiratory, and disability assessments using CareExchange in the home setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any form of Primary Immunodeficiency Disease
* Males and Females
* ≥ 15 and ≤ 85 years of age
* 5% treatment Naïve IVIg for the treatment of PIDD
* Ability to have Gammaplex® IVIg prescribed under the discretion of the patient's treating physician in accordance with standard treatment practices for the entire duration of the study
* Ability and willingness to provide informed consent and comply with study requirements and procedures
* Ability to read and write English
* Understanding of study procedures and ability to comply with study procedures for the entire length of the study
* Eligible for infusion services by AxelaCare Health Solutions, LLC, in collaboration with the subject's prescribing physician and insurance provider

Exclusion Criteria:

* The presence of any medical condition that the investigator and/or prescribing physician deems incompatible with participation in this trial.
* Prisoners, and other wards of the state
* Determined to have non-competency of data collection requirements (physical assessments and use of an iPAD™) by either the home infusion nurse and/or Caregiver.
* Receiving Subcutaneous Immunoglobulin (SCIg) Therapy during study participation.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and Females between 15-85 years of age with any form of PIDD who are considered 5% IVIg treatment naïve and whose physician has decided to prescribe Gammaplex® IVIg therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Analysis of collected data captured in CareExchange will demonstrate the ability to show and track changes in outcome data in 5% treatment naïve IVIg PIDD patients in the home setting. | 1 year

SECONDARY OUTCOMES:
Evaluate the profile physician usage (dose and timing) with Gammaplex®. | 1 year
Evaluate physician feedback to having real-time access to 5% treatment naïve IVIg PIDD data captured during home infusions. | 1 year
Evaluate the safety profile of using a 5% treatment naïve IVIg in PIDD patients in the home setting. | 1 year
Demonstration of response rate for those receiving IVIg therapies. | 1 year
Demonstration of changes in outcomes as a result of changes made in IVIg dose and frequency during study participation. | 1 year
Demonstration of measured variables within patients who receive IVIg therapies. | 1 year
Evaluate the effectiveness of whether CareExchange leads to better QOLs and overall patient reported outcomes. | 1 year
Other potential impacts on change in outcomes across patient demographics (age, sex, race, ethnicity, etc.). | 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hoag Medical Group (In Alliance with St. Joseph Heritage Healthcare), Newport Beach, California
  - IMMUNEOe International Research Centers, Centennial, Colorado
  - Atlanta ENT, Atlanta, Georgia
  - AxelaCare Health Solutions, LLC, Lenexa, Kansas